CLINICAL TRIAL: NCT07341776
Title: Evaluation of Emergency Medication in Children With Food Allergies: a Prospective, Randomized Clinical Multicenter Study Comparing Antihistamines Versus Antihistamines Plus Steroids in a Controlled Setting of Oral Food Challenges in Children.
Brief Title: Steroid Use in Treatment of Allergic Reactions to Food
Acronym: SAFARI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Trueck (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor-Investigator, Johannes Trueck, Head, Division of Allergy, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC-2025-00320; HumRes67580 (Registry Identifier: Humanforschung Schweiz); SNCTP000006696 (Registry Identifier: Humanforschung Schweiz)
Record Dates: First submitted 2025-12-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Anaphylactic Reaction; Anaphylaxis; Allergy in Children; IgE Mediated Food Allergy
MeSH Terms: conditions — Anaphylaxis; Food Hypersensitivity | interventions — Histamine Antagonists; Dimethindene; levocetirizine; Betamethasone; Prednisolone; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antihistamines plus oral steroids (Active Comparator): Participants receive oral antihistamines plus oral systemic corticosteroids for treatment of allergic reactions occurring during the oral food challenge. Intramuscular adrenaline may be administered as rescue medication if clinically indicated.
  Interventions: Drug: Antihistamines; Drug: Systemic corticosteroids; Drug: Adrenaline (rescue medication)
- Antihistamines only (no steroids) (Active Comparator): Participants receive oral antihistamines without systemic corticosteroids for treatment of allergic reactions occurring during the oral food challenge. Intramuscular adrenaline may be administered as rescue medication if clinically indicated.
  Interventions: Drug: Antihistamines; Drug: Adrenaline (rescue medication)

INTERVENTIONS:
Drug: Antihistamines — Oral administration of antihistamines for treatment of allergic symptoms during the oral food challenge.
  Other Names: Dimetindene maleate; Levocetirizine
Drug: Systemic corticosteroids — Oral administration of systemic corticosteroids as adjunctive treatment of allergic reactions during the oral food challenge.
  Other Names: Betamethasone; Prednisolone
  Arms: Antihistamines plus oral steroids
Drug: Adrenaline (rescue medication) — Intramuscular administration of adrenaline as rescue treatment for severe allergic reactions (anaphylaxis), administered as clinically indicated.
  Other Names: Adrenaline

SUMMARY:
In this study, the investigators want to find out whether a specific medication commonly used for severe allergic reactions is really necessary. When children have allergic reactions to foods, they are often given medications to relieve the symptoms. In addition to adrenaline and antihistamines, steroids are frequently administered in German-speaking Switzerland. However, it is unclear whether steroids are really helpful in this situation. To investigate this, the investigators are comparing two groups: one group receives additional steroids, and the other does not. Which treatment a participant receives is decided randomly, like flipping a coin. The study takes place during a pre-scheduled provocation test at the clinic. If an allergic reaction occurs, the usual emergency medications will be administered. Doctors will closely monitor how the reaction develops. No additional tests or visits are required. The results of this study could help improve allergy treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed IgE-mediated food allergy

Exclusion Criteria:

* Non-IgE mediated food allergies
* Non-food allergies
* Age outside the specified range
* Contraindications for an oral food challenge or oral steroid use within one week before the challenge.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to complete resolution of allergic symptoms | From onset of allergic symptoms during the oral food challenge until complete resolution of all allergic symptoms, assessed up to 24 hours.
  Time from onset of allergic symptoms during the oral food challenge until complete resolution of all allergic symptoms, comparing treatment with antihistamines alone versus antihistamines plus oral steroids.

SECONDARY OUTCOMES:
Total number of adrenaline doses and cumulative adrenaline dose | From onset of allergic reaction during the oral food challenge until resolution of symptoms or end of post-reaction observation period, assessed up to 24 hours.
  Total number of intramuscular adrenaline administrations and cumulative adrenaline dose administered per participant for treatment of allergic reactions during the oral food challenge.
Total number of antihistamine doses and cumulative antihistamine dose | From onset of allergic reaction during the oral food challenge until resolution of symptoms or end of post-reaction observation period, assessed up to 24 hours.
  Total number of oral antihistamine administrations and cumulative antihistamine dose administered per participant for treatment of allergic reactions during the oral food challenge.
Severity of allergic reaction | From onset of allergic reaction during the oral food challenge until resolution of symptoms or end of post-reaction observation period, assessed up to 24 hours.
  Severity of allergic reactions assessed using PRACTALL consensus definitions and documented on a standardized monitoring form during the oral food challenge.
Hospitalization and intensive care unit admission | From onset of allergic reaction during the oral food challenge until hospital discharge or end of observation period, assessed up to 24 hours.
  Occurrence of hospitalization or admission to an intensive care unit (ICU) for management of allergic reactions occurring during the oral food challenge.
Time from onset of allergic symptoms to patient discharge | From onset of allergic symptoms during the oral food challenge until patient discharge, assessed up to 24 hours.
  Time from onset of allergic symptoms leading to discontinuation of the oral food challenge until discharge from hospital or outpatient unit.
Late-phase allergic reactions | From resolution of initial allergic symptoms during the oral food challenge until 24 hours after onset of the allergic reaction.
  Occurrence of late-phase allergic reactions, defined as recurrence or worsening of allergic symptoms after complete resolution of the initial reaction, without further allergen exposure, following treatment during the oral food challenge.

OTHER OUTCOMES:
Adverse events | Up to 24 hours after onset of the allergic reaction.
  Frequency and severity of adverse events occurring after administration of study medications during the oral food challenge, categorized by type and severity according to standard adverse event definitions.
Rebound allergic symptoms | Up to 24 hours after onset of the allergic reaction.
  Occurrence of rebound allergic symptoms, defined as recurrence of allergic symptoms after initial complete resolution, without further allergen exposure, following treatment during the oral food challenge. Severity of rebound symptoms will be documented.
Additional medical interventions | Up to 24 hours after onset of the allergic reaction.
  Occurrence and type of additional medical interventions required after initial treatment of an allergic reaction during the oral food challenge, including repeat doses of antihistamines, administration of intramuscular adrenaline, or hospital admission.
Length of hospital stay and intensive care unit stay | Through hospital or ICU discharge (up to 24 hours after onset of the allergic reaction).
  Duration of hospital stay and, if applicable, ICU stay for participants admitted due to the allergic reaction during the oral food challenge; prolonged stays beyond the 24-hour assessment window will be recorded as adverse events/serious adverse events.
Prolonged observation period after allergic reaction | Up to 24 hours after onset of the allergic reaction.
  Proportion of participants requiring extended clinical observation due to persistent or worsening symptoms after initial treatment during the oral food challenge.
Patient and guardian assessment of symptom severity | Baseline and up to 24 hours after onset of the allergic reaction.
  Patient- and/or parent/guardian-reported assessment of symptom severity before and after onset of the allergic reaction during the oral food challenge. Symptom severity is assessed using standardized rating tools appropriate for age, including a face-based scale for children and a visual analogue scale (VAS-style) for parents/guardians.
Pollen exposure and weather conditions on the day of the oral food challenge | Day of the oral food challenge (Day 0).
  Documentation of ambient pollen exposure and weather conditions on the day of the oral food challenge, including pollen burden and relevant meteorological parameters, to allow exploratory assessment of their potential influence on allergic symptom severity and clinical course.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Children's Hospital Basel, Basel, Basel
  - University Children's Hospital, Zürich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Undecided